CLINICAL TRIAL: NCT00142532
Title: Acupuncture for Post-Thoracotomy Pain: A Randomized Controlled Trial
Brief Title: Acupuncture for Post-Thoracotomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Barrie Cassileth, PhD, Memorial Sloan Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-073
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer; Pain
Keywords: Acupuncture; Pain; Lung Cancer; Thoracotomy; Surgery
MeSH Terms: conditions — Lung Neoplasms; Pain | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): At the time of pre-op preparation, 18 semi-permanent intradermal acupuncture studs will be placed at acupuncture points in the back, two will be placed in the legs and two in the ear. All studs will be replaced when the epidural is removed or, for patients without epidurals, shortly before discharge. The new leg and auricular studs will then be removed at eleven days; the new back studs will be removed at the three week post-discharge consult.
  Interventions: Procedure: Acupuncture and Questionnaires
- 2 (Placebo Comparator): The treatment is the same as for the true acupuncture group, with the following exceptions. The studs in the back will be dummy studs have no needle and that have been used in previous research at MSKCC. The back studs will be placed halfway between the upper and lower border of spinous processes T2 to T10, approximately 0.5 cun (~1.25cm) from the spine. The leg studs will be placed at 2 cun (~5cm) posterior to GB34 on the posterior of the lower leg. No studs will be placed in the ear; rather studs will be placed on the anterior arm, 3 cun (~ 5cm) proximal and 3 cun (~ 5cm) medial to the midpoint of the antecubital crease.
  Numerical rating scale of pain; total opioid use; Medication Quantification Scale; length of stay; Brief Pain Inventory
  Interventions: Procedure: Placebo Acupuncture, Questionnaires

INTERVENTIONS:
Procedure: Acupuncture and Questionnaires — Acupuncture 30 day treatment BL12 - 19 and extra point Wei Guan Xia Shu Each side of the spine,1.5 cun (~2.5cm) lateral to the lower border of spinous process of the T2 - 10 spinal vertebrae respectively 4 weeks ST36, Below the knee, 3 cun (~7.5cm) inferior to the lower border of the patella, one finger breadth lateral to the anterior crest of the tibia. One week following removal of epidural.
  Shenmen, bilaterally. At the lateral 1/3 of the triangular fossa in the auricle.One week following removal of epidural.
  Questionnaires 30 / 60 / 90 Day and 12 Month Follow-up-Numerical rating scale of pain; total opioid use; Medication Quantification Scale; length of stay; Brief Pain Inventory
  Arms: 1
Procedure: Placebo Acupuncture, Questionnaires — The back studs will be placed halfway between the upper and lower border of spinous processes T2 to T10, approximately 0.5 cun (~1.25cm) from the spine. The leg studs will be placed at 2 cun (~5cm) posterior to GB34 on the posterior of the lower leg. No studs will be placed in the ear; rather studs will be placed on the anterior arm, 3 cun (~ 5cm) proximal and 3 cun (~ 5cm) medial to the midpoint of the antecubital crease.
  Pain will be assessed by a 0 - 10 point numerical rating scale (NRS) marked "no pain" at one end and "worst pain" at the other.
  Arms: 2

SUMMARY:
Pain after surgery for lung cancer (thoracotomy) may persist for years and require long-term analgesic use. Prior studies have shown that acupuncture reduces pain and medication use in the early post-operative period after abdominal surgery, suggesting that acupuncture may have a role in preventing chronic post-thoracotomy pain. This study is being done in order to determine the effects of acupuncture on pain in patients undergoing surgery for lung cancer.

DETAILED DESCRIPTION:
Rationale:

Acupuncture is the insertion of very fine needles into the skin to treat symptoms. In recent years, researchers have come to understand how acupuncture might work in terms of nerve stimulation and the release of chemical messages in the body. Researchers have found evidence that acupuncture is useful in treating a variety of conditions, including headache, nausea, and pain after surgery.

Pain is a common problem after surgery for lung cancer. Many patients experience pain in the first few days after surgery, despite medication. In some patients, this pain can last for many months or years afterwards.

Purpose:

A pilot study of acupuncture in patients undergoing lung cancer surgery was conducted previously and found that this study was feasible to implement and well-received by patients. We now wish to conduct a larger study in order to determine the effects of acupuncture on pain in patients undergoing surgery for lung cancer.

* To determine whether acupuncture versus placebo acupuncture after thoracotomy reduces pain or analgesic use
* To determine whether acupuncture affects the immediate post-operative period and/or 30, 60,90 days and approximately 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral thoracotomy at Memorial Sloan-Kettering Cancer Center (MSKCC)
* Age greater than or equal to 18 years old.

Exclusion Criteria:

* Any of the following procedures: hemiclamshell, clamshell, extrapleural approach, chest wall involvement, esophagectomy. These more extensive procedures have a higher risk of complications.
* Acupuncture treatment in the previous six weeks, to discount any persisting effect of acupuncture
* Platelets < 20,000 or International Normalized Ratio (INR) > 2.5 or absolute neutrophil count (ANC) < 0.5; though it would be unusual for any patient to be operated on with such values, it seems wise as a precautionary measure to avoid risk of bleeding from acupuncture.
* Known cardiac conditions constituting a high or moderate risk of endocarditis as defined by the American Heart Association criteria
* Patients unable to remove studs without assistance, who have no home assistance, and who are unable or unwilling to return to the hospital in the event that they decide to remove studs before the post-discharge visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine whether acupuncture versus placebo acupuncture after thoracotomy reduces pain or analgesic use | one year
To determine whether acupuncture affects the immediate post-operative period and/or 30, 60, 90 days and approximately 12 months later | one year

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Cassileth, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://mskcc.org